CLINICAL TRIAL: NCT00894296
Title: Magnetoencephalographic (MEG) Correlates of Negative Symptoms in Patients Suffering From Schizophrenia and Their Influence by Add-on Treatments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0027-08-SHA
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Schizophrenia
Keywords: MEG; schizophrenia; negative symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: schizophrenia patients
- 2: healthy control

SUMMARY:
The objective of the suggested study is to identify changes in MEG correlates caused by the add-on treatment with the changes in negative symptoms of schizophrenia by comparing the change in the MEG correlates of the subjects before and during usage of new add on treatments for negative symptoms.

The investigators hypothesize that the gravity of negative symptoms will correlate with a trend towards more aberrant electroencephalographic correlates mainly in continuous parameters, with an emphasis on alpha and delta bands

DETAILED DESCRIPTION:
There is a paucity of information regarding electrophysiological correlates of negative symptoms in patients suffering from schizophrenia. The proposed study is set out to compare the MEG correlates of negative symptoms in patients suffering from schizophrenia to those of healthy controls in terms of both relevant ERP components and quantified (continuous) MEG.

The presented study will include two parts: Part A will explore the electrophisological correlates of negative symptoms in patients suffering from schizophrenia using MEG. The study will do so by comparing the electrophisological correlates of schizophrenia patients suffering from negative symptoms and stable on psychiatric treatment to those of healthy controls. In the second part of the study data from part A of patients that have started new add-on treatments for negative symptoms will be compared to parallel data acquired after stabilization on the new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Study Group (Schizophrenia Patients) Inclusion Criteria
* Patients between the ages of 18-65 (male and female), Diagnosed in the past as suffering from schizophrenia. The diagnosis will be reaffirmed according to ICD criteria.
* Right hand dominant.
* Scores in PANSS negative questionnaire above 21 and positive symptom less than 24.
* Gave informed consent for participation in the study.
* Stable on the same antipsychotic medication for at least a month prior to entering the study Control Group (healthy Subjects)

Inclusion criteria:

* Healthy man and woman
* Ages 18-65
* Right handed

Exclusion Criteria:

* Study Group (Schizophrenia Patients) (To prevent MEG artifacts by non relevant electric interference or brain conditions)
* History of epilepsy, seizure, or hot spasm, sever head injuries.
* History of metal in the head (outside the mouth space).
* History of surgery including metal implant or history of metal particles in the eye, pacemaker, or any other medical pump.
* History of migraines.
* History of drug or alcohol abuse during the last year. Inability to achieve satisfying level of communication with the subject Control Group (healthy Subjects)
* History of psychiatric diagnosis
* Drug or alcohol addiction in the year prior to the study
* History of epilepsy, seizure, or hot spasm.
* History of head injuries.
* History of metal in the head (outside the mouth space).
* History of surgery including metal implant or history of metal particles in the eye, pacemaker, or any other medical pump.
* History of migraines.
* Use of psychotropic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: schizophrenia patients and healthy subjects between the ages 18-65
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures will include continuous and ERP (Event Related Potential) MEG (Magnetoencephalograph) data | four months

CONTACTS AND LOCATIONS:
Locations (1):
- Bar-Ilan University, Givat Shmuel, Israel